CLINICAL TRIAL: NCT01051505
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral AZD5069 After Administration of Multiple Ascending Doses for 8 Days in Healthy Male or Female Subjects
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Multiple Ascending Doses of AZD5069 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: D3550C00007
Record Dates: First submitted 2010-01-11; First posted 2010-01-18 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: Phase I; multiple ascending dose; Safety; Tolerability; Healthy Volunteer
MeSH Terms: interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD5069
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5069 — oral suspension dose of AZD5069. Multiple doses will be given once daily on day 1 and day 8 and twice daily on days 2 to 7
  Arms: 1
Drug: Placebo — oral suspension dose of matched placebo. Multiple doses will be given once daily on day 1 and day 8 and twice daily on days 2 to 7
  Arms: 2

SUMMARY:
The purpose of this study is to explore the safety and tolerability of AZD5069 at steady-state, following twice a day oral dosing in healthy subjects.

AZD5069 is being developed by AstraZeneca and this study is being carried out on behalf of the sponsor by Quintiles Drug Research Unit at Guy's Hospital, London. This is the second time that AZD5069 will be administered to humans in clinical trials. We are conducting this study to determine whether AZD5069 is safe and well tolerated by healthy males and females at different dose levels over an 8-day dosing period. We will also be studying how quickly AZD5069 is absorbed into and cleared by the body. It is planned that there will be up to 3 dose groups in the study and each group will consist of up to 12 volunteers, with 9 receiving the active drug and 3 receiving placebo. The study involves 3 visits over approximately 8 weeks, and will include 1 residential visit lasting 10 nights and a follow up.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent
* Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg
* Healthy male or female (of non child bearing potential)volunteers with suitable veins for cannulation or repeated venepuncture

Exclusion Criteria:

* Subjects must not have any clinically significant disease or disorder, which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results, or the subjects ability to participate
* Subjects must not have any history of gastrointestinal, liver or kidney disease, or any other condition known to interfere with how drugs are absorbed, used or eliminated by the body
* Subjects must not have had any significant illness or medical/surgical procedures or injuries with 4 weeks of administration of the investigational product

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Adverse events, electrocardiograms (ECGs), laboratory variables, blood pressure, pulse rate, body temperature, QT interval and continuous cardiac monitoring using telemetry | Baselines assessments at Visit 1 (enrolment) or pre-dose on Day 1 with assessments during Visit 2 at protocol defined time-points post-dose until 96hr post final dose. Follow up assessments at Visit 3

SECONDARY OUTCOMES:
Pharmacokinetic profile: concentration of AZD5069 in blood | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose
Assessment of ex vivo GROa stimulated CD11b expression on neutrophils in whole blood | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose
Measurement of the effect of AZD5069 on blood cells | Samples collected at Visit 2 from pre-dose and at regular protocol defined intervals up to 96 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, MBBS, DCPSA, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, London Bridge, United Kingdom

REFERENCES:
- [Derived] Cullberg M, Arfvidsson C, Larsson B, Malmgren A, Mitchell P, Wahlby Hamren U, Wray H. Pharmacokinetics of the Oral Selective CXCR2 Antagonist AZD5069: A Summary of Eight Phase I Studies in Healthy Volunteers. Drugs R D. 2018 Jun;18(2):149-159. doi: 10.1007/s40268-018-0236-x. PMID 29856004
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1337&filename=D3550C00007_Study_Synopsis.pdf